CLINICAL TRIAL: NCT07165587
Title: Venous Thromboembolism in Pelvic Ring and Acetabular Fractures - A Prospective Cohort Study
Brief Title: Incidence of Venous Thromboembolism in Patients With Pelvic and Acetabular Fractures (PAF)
Acronym: PAF-VTE
Status: Completed | Type: Observational
Sponsor: Department of Trauma and Reconstructive Surgery at Eberhard Karls University Tuebingen, BG Klinik Tu (Other)
Responsible Party: Sponsor
Other Study IDs: PAF-VTE
Record Dates: First submitted 2025-09-01; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Pelvic Fractures; Acetabular Fractures; Pelvic Trauma; Venous Thromboembolic Event; Venous Thromboembolism; Thromboprophylaxis; Pulmonary Embolism and Thrombosis
Keywords: observational study; pelvic fracuture; acetabular fracture; thromboprophylaxis; venous thromboembolic event
MeSH Terms: conditions — Hip Fractures; Venous Thromboembolism; Pulmonary Embolism; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with pelvic and/or acetabular fractures: Adult patients (≥18 years) admitted with pelvic, acetabular, or combined fractures. All participants receive standardized thromboprophylaxis with enoxaparin 4,000 IU twice daily as part of routine clinical care and undergo duplex ultrasound screening during hospitalization
  Interventions: Diagnostic Test: Bilateral duplex ultrasonography

INTERVENTIONS:
Diagnostic Test: Bilateral duplex ultrasonography — Bilateral duplex ultrasound screening performed during hospitalization to detect symptomatic and asymptomatic deep vein thrombosis in patients with pelvic and acetabular fractures.

SUMMARY:
The goal of this observational study is to investigate the incidence of venous thromboembolism (VTE) in patients with pelvic and acetabular fractures (PAF). The main question it aims to answer is:

What is the incidence of VTE in PAF patients receiving standardized thromboprophylaxis with enoxaparin 4,000 IU twice daily?

Participants admitted with a pelvic, acetabular, or combined fracture receive thromboprophylaxis as part of their routine clinical care. All participants undergo bilateral duplex ultrasound screening during hospitalization to detect both symptomatic and asymptomatic deep vein thrombosis. If pulmonary embolism is clinically suspected, computed tomography pulmonary angiography is performed.

The study aims to provide prospective observational data on VTE incidence and its association with fracture type, patient risk profile, and treatment modality.

DETAILED DESCRIPTION:
Pelvic and acetabular fractures (PAF) are serious injuries that carry a high risk of complications, including venous thromboembolism (VTE). VTE, which includes deep vein thrombosis (DVT) and pulmonary embolism (PE), is one of the most relevant and potentially life-threatening events in trauma patients. While VTE incidence in PAF patients has been reported to range widely in the literature, prospective data with standardized screening and prophylaxis are scarce.

This prospective observational cohort study investigates the incidence of VTE in adult patients admitted with pelvic, acetabular, or combined fractures. All participants receive standardized thromboprophylaxis with enoxaparin 4,000 IU administered twice daily, according to institutional protocol. In addition to routine clinical management, bilateral duplex ultrasonography is systematically performed during hospitalization to detect both symptomatic and asymptomatic DVT. In cases where pulmonary embolism is clinically suspected, computed tomography pulmonary angiography is carried out.

The primary outcome of the study is the incidence of VTE during the index hospital stay. Secondary outcomes include bleeding complications, and the association of fracture type, patient risk profile, and treatment modality with the occurrence of VTE.

The study is designed to provide high-quality observational data that will contribute to the understanding of VTE risk in this vulnerable patient population and may help inform future guidelines on thromboprophylaxis in pelvic and acetabular fracture care.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* Patients admitted with pelvic ring, acetabular, or combined pelvic-acetabular fracture
* Received thromboprophylaxis with enoxaparin 4,000 IU twice daily
* Hospital admission within the screening period
* Informed consent

Exclusion Criteria:

* Pathological fractures
* Thrombophilia
* Pre-existing oral anticoagulation
* Dementia
* Thromboprophylaxis other than enoxaparin 4,000 IU twice daily
* Admission outside the screening period
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) admitted to the BG Trauma Center at the University Hospital Tübingen with acute pelvic, acetabular, or combined pelvic-acetabular fractures. All participants received standardized thromboprophylaxis with enoxaparin 4,000 IU twice daily and underwent systematic duplex ultrasound screening during hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of venous thromboembolism (VTE) during hospital stay | Conservative: 48h, days 3-6 post-trauma. Operative: ≤48h post-trauma, postop days 2-5. Baseline only if admitted ≤48h. Additional exams if clinical suspicion of VTE during hospitalization.
  Detection of symptomatic and asymptomatic VTE (deep vein thrombosis or pulmonary embolism) during index hospitalization, assessed by routine duplex ultrasound and clinical imaging.

SECONDARY OUTCOMES:
Bleeding complications | From admission until hospital discharge (up to 60 days); bleeding events were continuously monitored throughout the entire index hospitalization.
  Number of bleeding events related to thromboprophylaxis
Association of VTE with fracture type and treatment modality | VTE assessed during index hospitalization: conservative patients at 48h and days 3-6 post-trauma; operative patients at ≤48h post-trauma and postop days 2-5; additional exams if clinical suspicion, until discharge (up to 60 days).
  Exploratory analysis of VTE incidence according to pelvic vs. acetabular vs. combined fractures and operative vs. non-operative treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Trauma and Reconstructive Surgery, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) underlying the results reported in this study will not be made publicly available due to local data protection regulations. Summary-level results will be shared in publications and upon reasonable request to the corresponding author.

REFERENCES:
- [Background] Mahmoud SS, Esser M, Jain A. Thromboembolic events in pelvic and acetabulum fractures: a systematic review of the current literature on incidence, screening, and thromboprophylaxis. Int Orthop. 2022 Aug;46(8):1707-1720. doi: 10.1007/s00264-022-05431-z. Epub 2022 May 11. PMID 35543748
- [Background] Wang P, Kandemir U, Zhang B, Wang B, Li J, Zhuang Y, Wang H, Zhang H, Liu P, Zhang K. Incidence and Risk Factors of Deep Vein Thrombosis in Patients With Pelvic and Acetabular Fractures. Clin Appl Thromb Hemost. 2019 Jan-Dec;25:1076029619845066. doi: 10.1177/1076029619845066. PMID 31014089
- [Background] Zhao W, Zhao J, Liu T, Liu Z, Liu L, Zhang Y. Incidence and risk factors of preoperative deep venous thrombosis following pelvic and acetabular fractures: a retrospective case-control study. J Orthop Surg Res. 2022 Feb 5;17(1):77. doi: 10.1186/s13018-022-02972-2. PMID 35123537